CLINICAL TRIAL: NCT05433064
Title: Spinal Cord Stimulation for Spinal Cord Injury Patients - Regain Walk and Alleviate Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCMF-EP 110-02(111)
Record Dates: First submitted 2022-04-17; First posted 2022-06-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Epidural Stimulator (Experimental): Subjects will be implanted with 16-electrode epidural array in the T11-L1 area of the spinal cord. After 2 weeks recovery,patients will undergo a structured program of physical rehabilitation and electrical stimulation.
  Interventions: Device: Epidural Stimulator

INTERVENTIONS:
Device: Epidural Stimulator — Subjects will be implanted with 16-electrode epidural array in the T11-L1 area of the spinal cord. After 2 weeks recovery,patients will undergo a structured program of physical rehabilitation and electrical stimulation.
  Other Names: Abbott Lead-3219

SUMMARY:
The study aims to examine the plausible interventional mechanisms underlying the effects of epidural spinal cord stimulation.

DETAILED DESCRIPTION:
The purpose of this study is for the treatment of spinal cord injury (SCI) paralysis patients use the signal by electrophysiological analysis of epidural spinal cord stimulation (SCS) settings that promote lower limb activity so that SCI patients can restore the ability to stand and walk under multiple sensory stimuli and multimodal electrical stimulation rehabilitation. The investigators hope to establish an atresia nerve regulation strategy and observe that the original blocked neural circuits can improve nerve plasticity by SCS. Even can establish new connections through residual nerves and allow SCI patients to rebuild neural circuits without SCS to restore lower limb mobility and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* SCI ASIA: A, B, C,D
* Between 20 and 70 year of age
* >1 year post SCI
* Complete or incomplete spinal cord injury.
* Expected will undergo spinal cord stimulation surgery.
* Continued rehabilitation after surgery for spinal cord injury.
* Able to comply with procedures and follow up.
* Stable medical condition without cardiopulmonary disease or dysautonomia that would contraindicate participation in lower extremity rehabilitation or testing activities

Exclusion Criteria:

* Have significant cognitive impairment (MMSE<24).
* Had a mental illness within one year or been treated in the past.
* Have Major depressive disorder.
* Active cancer diagnosis.
* Painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore, or urinary tract infection that might interfere with stand or step training.
* Cardiovascular or musculoskeletal disease or injury that would prevent full participation in physical therapy intervention.
* Unable to read and/or comprehend the consent form.
* Have concerns about this trial and do not sign consent.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
6-Meter Time Up and Go (6TUG) | To measure assessing change between pre-implant and every 3 months until 24 months.
  To evaluate gait for subjects who can walk by assistive device or independently.
Assessment of volitional movement of lower limbs using electromyographic analysis | To measure assessing change between pre-implant and every 3 months until 24 months.
  Average of 6-repetitive EMG activity for each superficial component of muscles from a five-second ramp contraction to the end of a ten-second rest
Trunk stability measurement (trunk control assessment) | To measure assessing change between pre-implant and every 3 months until 24 months.]
  To assess the sitting and walking dynamic balance by displacing the center of pressure (CoP) from the force plate and the trunk accelerations with a tri-axial accelerometer. The experiment includes sitting and walking.pressure (CoP) from the force plate and the trunk accelerations with tri-axial accelerometer.

SECONDARY OUTCOMES:
Change in Quality of Life (QOL) as measured by the World Health Organization Quality of Life (WHOQOL-BREF) | Baseline; at 1 - 4 - 7 - 13 - 19 - 25 months after implantation
  The WHOQOL-BREF is a self-administered questionnaire comprising 26 questions on the individual's perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely". , The higher the score, the better the quality of life
Change in spasticity as measured by the Modified Ashworth Scale (MAS) | Baseline; at 1 - 4 - 7 - 13 - 19 - 25 months after the implantation
  It is mainly used to assess muscle spasm (spasticity). The muscle tension is divided into 0-4 grades. The lower the score, the closer to normal. The higher the score, the more severe the spasticity.
Change in motor recovery as measured by the Total American Spinal Injury Association (ASIA) motor score | Baseline; at 1 - 4 - 7 - 13 - 19 - 25 months after implantation
  The American Spinal Injury Association (ASIA) Standard Neurological Classification of Spinal Cord Injury is a standard method of assessing the neurological status, including motor and sensory evaluations, of a person who has sustained a spinal cord injury.
Change in ability (or inability) to safely balance as measured by the Berg Balance Scale (BBS) | Baseline; 7 months after implant
  It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.a 14-item scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Tzung Tsai, M.D., Ph.D., Principal Investigator — Hualien Tzu Chi General Hospital
Locations (1):
- Buddhist Tzu Chi Medical Foundation Hualien Tzu Chi Hospital, Hualien City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu MY, Chen LH, Yang CH, Wu CC, Huang XL, Yan LC, Lin SZ, Wang PK, Lee CH, Chen YC, Tsai ST. Synergistic effect of epidural electrical stimulation and exoskeleton walk training on dynamic balance for participants with spinal cord injury. J Spinal Cord Med. 2025 Oct 24:1-10. doi: 10.1080/10790268.2025.2574134. Online ahead of print. PMID 41134059
- [Derived] Chen YC, Huang XL, Cheng HY, Wu CC, Wu MY, Yan LC, Chen SY, Tsai ST, Lin SZ. Role of Epidural Electrode Stimulation in Three Patients with Incomplete AIS D Spinal Cord Injury. Biomedicines. 2025 Jan 10;13(1):155. doi: 10.3390/biomedicines13010155. PMID 39857740